CLINICAL TRIAL: NCT02059330
Title: A Phase 1, Open Label Study To Investigate The Effect Of Dose And Ethnicity On Palbociclib (PD-0332991) Pharmacokinetics In Japanese Healthy Volunteers
Brief Title: A Study To Investigate Palbociclib (PD-0332991) Pharmacokinetics In Healthy Subjects Of Japanese Descent Relative To Healthy Non-Asian Subjects, And To Determine If Changes In Palbociclib Dose Result In Proportional Changes In Palbociclib Plasma Exposure In Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: A5481032
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: Japanese PK-Bridging Study; dose-proportionality study; Palbociclib; PD-0332991; healthy volunteers
MeSH Terms: interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Subjects of Japanese Descent (Experimental): Enrolled Japanese subjects will receive four palbociclib single doses of differing dose amounts in fixed sequence over four treatment periods.
  Interventions: Drug: Palbociclib 75mg; Drug: Palbociclib 125mg; Drug: Palbociclib 100mg; Drug: Palbociclib
- Healthy Non-Asian Subjects (Experimental): Enrolled healthy non-Asian subjects will receive a single 125mg oral dose of palbociclib in a single treatment period.
  Interventions: Drug: Palbociclib 125mg

INTERVENTIONS:
Drug: Palbociclib 75mg — In Period 1, Japanese subjects will receive a single oral 75mg dose of palbociclib with food. Serial PK assessments will be collected over the next 120 hours.
  Other Names: PD-0332991
  Arms: Healthy Subjects of Japanese Descent
Drug: Palbociclib 125mg — In Period 2, Japanese subjects will receive a single oral 125mg dose of palbociclib with food. Serial PK assessments will be collected over the next 120 hours.
  Other Names: PD-0332991
  Arms: Healthy Subjects of Japanese Descent
Drug: Palbociclib 100mg — In Period 3, Japanese subjects will receive a single oral 100mg dose of palbociclib with food. Serial PK assessments will be collected over the next 120 hours.
  Other Names: PD-0332991
  Arms: Healthy Subjects of Japanese Descent
Drug: Palbociclib — In Period 4, Japanese subjects will receive a single oral dose of palbociclib with food. Serial PK assessments will be collected over the next 120 hours. The amount of the dose will be determined based on an interim analysis of the PK data from Periods 1 and 2.
  Other Names: PD-0332991
  Arms: Healthy Subjects of Japanese Descent
Drug: Palbociclib 125mg — In Period 1, healthy non-Asian subjects will receive a single oral 125mg dose of palbociclib with food. Serial PK assessments will be collected over the next 120 hours.
  Other Names: PD-0332991
  Arms: Healthy Non-Asian Subjects

SUMMARY:
This study will investigate the dose-proportionality of palbociclib pharmacokinetics in healthy subjects of Japanese descent. Approximately fourteen healthy Japanese subjects will receive four single doses of palbociclib (PD-0332991) with a minimum washout of 10 days between doses. Additionally, this study will investigate the effect of Japanese ethnicity of palbociclib pharmacokinetics by comparing palbociclib pharmacokinetics at a single dose-level between healthy subjects of Japanese descent and approximately fourteen healthy non-Asian subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be a healthy male or female of non-childbearing potential
* Subjects must have a BMI (Body Mass Index) between 17.5 and 30.5 kg/m2
* To be eligible for the Japanese cohort, subjects must have 4 biological grandparents who are Japanese that were born in Japan

Exclusion Criteria:

* Any condition affecting drug absorption (eg gastrectomy, achlorhydria, etc)
* Use of prescription or non-prescription drugs
* A QTc-interval >450msec or a QRS interval >120msec
* Pregnant or breastfeeding females, females of childbearing potential, and males who are unwilling or unable to use an effective method of contraception for the duration of the study and for 90 days after the last dose of palbociclib in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 0-120 hours
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Dose-normalised Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 0-120 hours
  AUC (0 - 8)DN= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8) divided by dose. It is obtained from AUC (0 - t) plus AUC (t - 8) all divided by the administered dose.
Maximum Observed Plasma Concentration (Cmax) | 0-120 hours
Dose-Normalised Maximum Observed Plasma Concentration (Cmax) | 0-120 hours

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0-120 hours
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Dose-Normalized Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0-120 hours
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast), all divided by the administered dose.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0-120 hours
Plasma Decay Half-Life (t1/2) | 0-120 hours
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Apparent Oral Clearance (CL/F) | 0-120 hours
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) | 0-120 hours
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481032&StudyName=A%20Study%20To%20Investigate%20Palbociclib%20%28PD-0332991%29%20Pharmacokinetics%20In%20Healthy%20Subjects%20Of%20Japanese%20Descent%20Relative%20To%20Healthy%20Non-Asian%20S